CLINICAL TRIAL: NCT03823092
Title: Polarization Perception in Health and Disease. Testing a New Sight Test: The TaNSiT Study
Brief Title: Polarization Perception in Health and Disease. Testing a New Sight Test
Acronym: TaNSiT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Warwickshire NHS Foundation Trust (Other)
Collaborators: Aston University (Other)
Responsible Party: Principal Investigator, Gary Misson, Consultant ophthalmologist, South Warwickshire NHS Foundation Trust
Other Study IDs: 17/WA/0180
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Cataract; Age Related Macular Degeneration; Pseudophakia; Macular Disease; Diabetic Retinopathy; Retinal Disease
Keywords: macular function; polarization perception; Haidinger's brush; vision testing; cataract; age related macular degeneration; pseudophakia; macular disease; retinal disease
MeSH Terms: conditions — Cataract; Macular Degeneration; Pseudophakia; Diabetic Retinopathy; Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Normal: phakic participants with no evidence of eye disorders
  Interventions: Diagnostic Test: polarization sensitivity
- Cataract: participants with cataract
  Interventions: Diagnostic Test: polarization sensitivity
- AMD: participants with age related macular degeneration
  Interventions: Diagnostic Test: polarization sensitivity
- Pseudophakic: particpiants who have had cataract surgery with intraocular lens implant
  Interventions: Diagnostic Test: polarization sensitivity
- other macula: participants with macular ddisorders other than AMD
  Interventions: Diagnostic Test: polarization sensitivity
- DR: participants with diabetic retinopathy
  Interventions: Diagnostic Test: polarization sensitivity

INTERVENTIONS:
Diagnostic Test: polarization sensitivity — test of polarization vision as described in Study Description

SUMMARY:
A study to assess the utility of human polarization pattern perception for the detection, diagnosis and monitoring of eye disease

DETAILED DESCRIPTION:
The recently described high sensitivity of the human eye to differentiate small angular differences in linear polarization and evidence supporting its macular origin (Misson, Anderson; 2017) suggests that human polarization sensitivity might be a useful diagnostic tool for macular disease. This augments a previous study in which we demonstrated the ability of the human visual system to detect isochromatic isoluminant polarization modulated pattern stimuli (Misson et al 2015).

This is an exploratory 'proof-of-concept' study to determine the clinical value of polarization pattern perception, PPP, in health and disease. We further propose that PPP might be valuable for the diagnosis, monitoring and early detection of macular disease. The latter includes common blinding conditions such as age related macular degeneration and diabetic retinopathy. It is also intended to investigate the effect of cataracts and cataract surgery on PPP: cataract surgery modifies the optics of the eye so might also modify PPP.

PPP is measured using a modification of the methodology described in (Misson et al 2015) and (Misson, Anderson; 2017) whereby polarization modulated patterns are presented on a modified LCD display. The observer's task is to report if they see an image and to describe the image. Images comprise simple patterns or traditional optotypes. A standard set of images are presented in pseudorandom order and the response recorded. A total score, the polarization pattern perception score PPP is then determined from the number of images seen/identified. A more refined metric, the polarization visual acuity pVA, will be derived from the response to the optotype stimuli. These data are then compared to conventional tests of visual structure and function including logMAR visual acuity, ocular examination and OCT scan data.

The study in anticipated to comprise:

Phase 1. Normative Evaluation: observational prospective cross-sectional.. A preliminary normative study will be undertaken on staff members. The aim is to quantify normative values in preparation for the clinical studies.

Hypotheses to be tested:

1. that healthy subjects can perceive polarization stimuli
2. that there is a threshold of polarization image resolution (pVA) analogous to visual acuity. Normative PPP and pVA data will be collected.

Phase 2 Patient Group: observational Prospective cross-sectional / case-control.

Phase 2 subjects will comprise normals and patients with cataracts/pseudophakia and/or AMD, other macular pathology, diabetic retinopathy..

The aim of this phase is to determine the effect, if any, of particular eye conditions on pVA/PPP alone and in comparison with other test parameters.

Hypotheses to be tested:

1. that eye conditions affect pVA/PPP
2. that specific eye conditions have a selective effect on pVA/PPP
3. that pseudophakia affects pVA/PPP

Phase 3: Cataract pre-op v post op pVA/PPP: prospective interventional case-control.

Timescale:concurrent with Phase 2 A subset of the phase 2 cataract patients will undergo cataract surgery according to clinical need. These patients are routinely reviewed 4 - 8 weeks post-op when the opportunity will arise to repeat pVA/PPP measurement. The fellow eye will serve as a control / provide data for repeatability assessment.

The aims of this phase are

1. to determine the repeatability of pVA/PPP testing in a heterogeneous patient group
2. to determine the effect of cataract surgery on the pre-operative pVA/PPP results
3. to determine if pVA/PPP is a useful determinant of post-operative visual outcome.

Hypotheses:

1. that pVA/PPP testing is repeatable
2. that there is a difference in pVA/PPP pre and post cataract surgery

ELIGIBILITY:
Inclusion Criteria:

- willing and able to provide informed consent

Exclusion Criteria:

* unwilling or unable to provide informed consent
* individuals wishing to exit the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and staff of the Eye Department of South Warwickshire NHS Trust
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
polarization sensitivity | 18 month
  determine and compare polarization sensitivity between groups

CONTACTS AND LOCATIONS:
Locations (1):
- South Warwickshire NHS Foundation Trust, Warwick, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Misson GP, Timmerman BH, Bryanston-Cross PJ. Human perception of visual stimuli modulated by direction of linear polarization. Vision Res. 2015 Oct;115(Pt A):48-57. doi: 10.1016/j.visres.2015.08.004. Epub 2015 Aug 28. PMID 26291073
- [Result] Misson GP, Anderson SJ. The spectral, spatial and contrast sensitivity of human polarization pattern perception. Sci Rep. 2017 Nov 29;7(1):16571. doi: 10.1038/s41598-017-16873-6. PMID 29185499